CLINICAL TRIAL: NCT03745573
Title: Preventing Violence Against Children in Schools: Protocol for a Cluster Randomised Controlled Trial of the EmpaTeach Behavioural Intervention in Nyarugusu Refugee Camp
Brief Title: Preventing Violence Against Children in Schools Study
Acronym: PVACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Institutes of Medical Research, Tanzania (Unknown); Innovations for Poverty Action, Tanzania (Unknown); International Rescue Committee (Other); Behavioural Insights Team (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11106
Record Dates: First submitted 2018-11-06; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Violence, Physical; Violence; Child Abuse; Violence Against Children
Keywords: corporal punishment, teacher violence, school violence, sexual violence

STUDY DESIGN:
Intervention Model Description: Schools will be randomised to receive the intervention or a wait-list control condition. Assignment will be parallel.
Masking Description: Due to the behavioural nature of the intervention, it is not possible to mask allocation to participants. Outcome assessors will not be told of allocation, but due to the nature of the intervention they should be assumed to be unmasked. The statistician performing the main trial analyses related to primary and secondary outcomes will be masked to allocation, but other investigators will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empateach Intervention (Experimental): All teachers in intervention schools will be invited to participate. Participants in the intervention condition will receive Empateach, a 10-week group intervention. Groups meet 14 times for 1-1.5 hour length sessions, which are led by peers. The aim of the Empateach intervention is to improve 'student and teacher well-being; self-regulation; teacher classroom management and teacher's use of positive discipline techniques. The intervention uses cognitive behavioural therapy techniques to change negative thought and behaviour patterns related to corporal punishment. The teachers receive information on alternatives to corporal punishment, planning exercises and reinforcement SMS, and because the intervention is in a group setting, social support to change their behaviours. They discuss their experiences and challenges in group sessions.
  Interventions: Behavioral: Empateach
- Wait-list control (No Intervention): Teachers in wait-list control schools will receive no specific interventions related to violence prevention during the study, but will receive the intervention after the study is over if it is shown to be effective (pending donor funding).

INTERVENTIONS:
Behavioral: Empateach — Empateach is a behavioural intervention for teachers.
  Arms: Empateach Intervention

SUMMARY:
To date, no interventions to prevent violence in refugee camp schools have ever been rigorously evaluated. The primary objective of this project is to test the effectiveness of the Empateach intervention to prevent physical violence from teachers to students in Nyarugusu Refugee Camp, Tanzania. Secondary objectives are to assess the impact of the Empateach intervention on student's depressive symptoms, experience of emotional violence and educational test scores. A two arm cluster RCT with parallel assignment will be conducted.

DETAILED DESCRIPTION:
School is one of the most common settings where children may experience violence; and emerging evidence suggests that in some settings, school staff may be one of the most common perpetrator of violence against children.To date, no interventions to prevent violence in refugee camp schools have ever been rigorously evaluated. The primary objective of this project is to test the effectiveness of the Empateach intervention to prevent physical violence from teachers to students in Nyarugusu Refugee Camp, Tanzania. Secondary objectives are to assess the impact of the Empateach intervention on student's depressive symptoms, experience of emotional violence and educational test scores.

The aim of the Empateach intervention is to improve 'student and teacher well-being; self-regulation; teacher classroom management and teacher's use of positive discipline techniques'. Participants in the intervention condition will receive a 10-week group intervention.

A two arm cluster RCT will be conducted, with parallel assignment and an approximately 1:1 allocation ratio. Cross-sectional surveys of students will be conducted at three time points: a baseline, a midline immediately after the 10 week intervention; and an endline 6 months after then end of the intervention. The primary outcome, violence from school staff to students, will be measured using an adapted version of the ICAST-CI.

ELIGIBILITY:
Inclusion Criteria:

* At the school level, all 27 primary and secondary schools in Nyarugusu refugee camp in Tanzania, will be eligible. The intervention is delivered to individual teachers, and all teachers working in included schools will be eligible to receive the intervention. The hypothesized intervention effect will be in all students being taught by participating teachers; however we will measure effects of the intervention in students who are aged 9 years and over. Data will be collected from both students and teachers.
* At the level of individual students, all students who can speak Kirundi or Swahili, and who are capable of providing assent, will be eligible to participate
* At the level of individual teachers, all teachers who can speak Kirundi or Swahili, and who are capable of providing informed consent, will be eligible to participate

Exclusion Criteria:

* there are no exclusion criteria at the School level
* for individual students, those who cannot speak Kirundi or Swahili, or who are not capable of providing assent
* for individual teachers, those who cannot speak Kirundi or Swahili, or who are not capable of providing informed consent

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2120 (Estimated)
Dates: Start 2018-11-16 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
physical violence | Assessed at 10-week follow-up
  students' self-reports of physical violence from school staff in the past week, as measured by a modified ICAST-CI

SECONDARY OUTCOMES:
physical violence | Assessed at 6-month follow-up
  students' self-reports of physical violence from school staff in the past week, as measured by a modified ICAST-CI
emotional violence | past 1 week; assessed at 10-week and 6-month follow-up
  students' self-reports of emotional violence from school staff, as measured by a modified ICAST-CI
depressive symptoms | past 2 weeks; assessed at 10-week and 6-month follow-up
  students' self-reports of emotional violence from school staff, as measured by a modified ICAST-CI
educational performance | assessed at the end of the school year, about 11-12 months from baseline
  test scores on yearly exams

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Devries, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine

IPD SHARING:
Plan to Share IPD: Undecided
We will explore making anonymised data available after the end of the study, subject to UK and Tanzanian regulations.

REFERENCES:
- [Derived] Bakari M, Shayo EH, Barongo V, Kiwale Z, Fabbri C, Turner E, Eldred E, Mubyazi GM, Rodrigues K, Devries K. Qualitative process evaluation of the EmpaTeach intervention to reduce teacher violence in schools in Nyarugusu Refugee Camp, Tanzania. BMJ Open. 2023 Sep 21;13(9):e069993. doi: 10.1136/bmjopen-2022-069993. PMID 37734883
- [Derived] Fabbri C, Rodrigues K, Leurent B, Allen E, Qiu M, Zuakulu M, Nombo D, Kaemingk M, De Filippo A, Torrats-Espinosa G, Shayo E, Barongo V, Greco G, Tol W, Devries KM. The EmpaTeach intervention for reducing physical violence from teachers to students in Nyarugusu Refugee Camp: A cluster-randomised controlled trial. PLoS Med. 2021 Oct 4;18(10):e1003808. doi: 10.1371/journal.pmed.1003808. eCollection 2021 Oct. PMID 34606500
- [Derived] Devries KM, Fabbri C, Allen E, Barongo V, Shayo E, Greco G, Kaemingk M, Qiu M, Steinacher R, Tol W, Rodrigues K. Preventing violence against children in schools (PVACS): protocol for a cluster randomised controlled trial of the EmpaTeach behavioural intervention in Nyarugusu refugee camp. BMC Public Health. 2019 Oct 15;19(1):1295. doi: 10.1186/s12889-019-7627-y. PMID 31615467